CLINICAL TRIAL: NCT02444286
Title: Observational Study of Heart Failure Patients With Clinically Significant Functional Mitral Regurgitation - Follow Up of the Former Participants in the RESHAPE-HF Trial (Abbott Vascular).
Brief Title: The RESHAPE-HF1-FU Study
Status: Withdrawn | Type: Observational
Why Stopped: study did never start, may be deleted from clinicaltrials.gov if possible
Sponsor: Institut fuer anwendungsorientierte Forschung und klinische Studien GmbH (Other)
Collaborators: University Medical Center Goettingen (Other)
Responsible Party: Sponsor
Other Study IDs: Version No. 1.0
Record Dates: First submitted 2015-05-12; First posted 2015-05-14 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2019-01

CONDITIONS: Mitral Valve Insufficiency
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- standard care group: optimal standard of care therapy
- device group: Follow-up of MitraClip device implantation plus optimal standard of care therapy

SUMMARY:
To evaluate the safety and efficiency of the MitraClip system in the treatment of patients with clinically significant mitral regurgitation with New York Heart Association (NYHA) Functional Class II to IV chronic heart failure.

DETAILED DESCRIPTION:
The purpose of the RESHAPE-HF1-FU Study is to follow up the safety and effectiveness of the MitraClip System in the treatment of clinically significant Functional Mitral Regurgitation (FMR) in patients with New York Heart Association (NYHA) Functional Class III or IV chronic heart failure, former participants in the RESHAPE-HF Trial (Abbott Vascular).

ELIGIBILITY:
Inclusion Criteria:

* Former participant in the RESHAPE-HF Trial (Abbott Vascular)
* Subject agrees to return for all required follow-up visits
* The subject has been informed of the nature of the study and agrees to the study's provisions and has provided written informed consent as approved by the respective clinical site's Ethics Committee

Exclusion Criteria:

* Withdrawal of Informed Consent
* Subject belongs to a vulnerable population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The RESHAPE- HF1-FU Study is an observational, multi-center clinical evaluation (follow-up) of the MitraClip device plus optimal standard of care therapy (subjects with Device) compared to optimal standard of care therapy alone (other subjects), of former participants in the RESHAPE-HF Trial (Abbott Vascular).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Estimated); Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
cardiovascular (CV) death | 24 months
  Composite rate of recurrent heart failure hospitalizations and cardiovascular (CV) death

SECONDARY OUTCOMES:
Mitral Regurgitation (MR) severity reduction | at 12 and 24 months
  Mitral Regurgitation (MR) severity reduction to mild or mild-to-moderate at 12 and 24 months
6 Minute Walk Test (6MWT) | at 6, 12 and 24 months
  Change in 6 Minute Walk Test (6MWT) distance at 6, 12 and 24 months over baseline
CV hospitalizations and CV death | 24 months
  Rate of recurrent CV hospitalizations and CV death
Quality of Life (QoL) | 12 months
  Change in Quality of Life (QoL) overall score, as measured by Kansas City Cardiomyopathy Questionnaire (KCCQ) at 12 months over baseline
New York Heart Association (NYHA) Functional Class | 6, 12 and 24 months
  Change in New York Heart Association (NYHA) Functional Class over baseline and proportions of patients in NYHA Functional Class I/II at 6, 12 and 24 months
Patient-reported Global Assessment (PGA) | 6, 12 and 24 months.
  Change in Patient-reported Global Assessment (PGA) of well-being at 6, 12 and 24 months

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Medical Center Goettingen, Göttingen
  - University Hospital Mainz, Mainz